CLINICAL TRIAL: NCT01802697
Title: A Phase i Single Center Study to Evalute the Safety, Tolerability and Pharmacokinetics of Intravenous IdeS After Administration of Single Ascending Doses in Healthy Male Subjects
Brief Title: Safety Study on IdeS in Healthy Volounteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 11-HMedIdeS-01; 2012-000969-21 (EudraCT Number)
Record Dates: First submitted 2013-02-27; First posted 2013-03-01 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
Keywords: volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IdeS (Experimental): Intravenous infusion
  Interventions: Drug: IdeS
- PBS Buffer (Placebo Comparator): Intravenous infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: IdeS
  Arms: IdeS
Drug: Placebo
  Arms: PBS Buffer

SUMMARY:
This is a first in man study to assess safety and tolerability of the IgG cleaving enzyme Immunoglobuli G degrading enzyme of streptococcus pyogenes (IdeS).

DETAILED DESCRIPTION:
A phase I study (11-HMedIdeS-01, EudraCT no. 2012-000 969-21) first in man single ascending dose study in 29 healthy subjects to investigate if IdeS is safe and well tolerated in doses up to 0.24 mg/kg body weight (BW).

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and sign informed consent
* BMI 19-30

Exclusion Criteria:

* Clinically significant disease
* Positive HIV, hepatistis B or C

  * Drug abuse
* Smoking
* Use of medication except paracetamol

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2013-02; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Safety as measured by adverse events | 64 days

SECONDARY OUTCOMES:
Peak plasma concentration of IdeS | 7 days

OTHER OUTCOMES:
Total IgG concentration | 64 days

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Malmqvist, MD, PhD, Principal Investigator — Clinical Trial Unit, SUS, Lund, Sweden
Locations (1):
- Clinical Trial Unit, FoU centrum Skåne, Skåne University hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Winstedt L, Jarnum S, Nordahl EA, Olsson A, Runstrom A, Bockermann R, Karlsson C, Malmstrom J, Palmgren GS, Malmqvist U, Bjorck L, Kjellman C. Complete Removal of Extracellular IgG Antibodies in a Randomized Dose-Escalation Phase I Study with the Bacterial Enzyme IdeS--A Novel Therapeutic Opportunity. PLoS One. 2015 Jul 15;10(7):e0132011. doi: 10.1371/journal.pone.0132011. eCollection 2015. PMID 26177518